CLINICAL TRIAL: NCT00221871
Title: Proper Dosage of Intravenous Ketamine When Used as an Adjuvant to Lidocaine in Intravenous Regional Anesthesia (IVRA).
Brief Title: Proper Dosage of Ketamine in Intravenous Regional Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHN02-0233-A
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2005-09

CONDITIONS: Pain.
MeSH Terms: conditions — Pain

INTERVENTIONS:
Drug: Different dosages of Ketamine

SUMMARY:
Ketamine added to Lidocaine can increase duration of pain relief following intraveonous regional anesthesia (IVRA). The purpose of this dose response study is to determine the minimum effective dosage of intravenous Ketamine, added to 3 mg/kg of Lidocaine. We anticipate that one dosage will provide us with the proper balance between sufficient anesthesia and minimal side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70
2. Weight: 50-100 kg
3. ASA: I, II, III
4. Carpal tunnel syndrome surgery, tenolysis, ganglion removal or any peripheral hand surgery that can be done by IVRA.

Exclusion Criteria:

1. Contraindication to IVRA such as sickle cell disease.
2. Any known hypersensitivity reaction to Ketamine.
3. History of chronic pain or regular medication with analgesics.
4. History of opioid dependence.
5. Drug of alcohol abuse.
6. Psychiatric disorder.
7. Allergy to acetaminophen or codeine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Colin McCartney, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada